CLINICAL TRIAL: NCT02794831
Title: Exposure to NSAIDs (Non Steroidal Anti-Inflammatory Drugs) and Severity of Community-acquired Bacterial Infections
Acronym: ANAIG
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Tours (Other); University Hospital, Grenoble (Other); Central Hospital, Nancy, France (Other); University Hospital, Limoges (Other); LA ROCHE SUR YON HOSPITAL (Unknown); Agence Nationale de sécurité du Médicament (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0364
Record Dates: First submitted 2016-05-11; First posted 2016-06-09 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Bacterial Infection
Keywords: NSAIDs; Bacterial Infections; Severity; Self Medication
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patient: Adult patient hospitalized in MCO in one of the study centers for severe community bacterial infection, infected with more than one site, and / or abscess collection, and / or a per-cutaneous drainage of the infection, and / or septic surgery.
- control: Patient hospitalized in the same center (different service or not), during the week or months of the inclusion of cases for infection without abscess or invasive procedure, only one infected site

SUMMARY:
* NSAIDs are widely consumed, and some are currently available for self-medication with indications 'Pain and Fever' (Cavalié, National Agency for Drug Safety (ANSM), 2014)
* There is no recommendation to limit their use in bacterial infections except for chicken pox in children.
* To date, no study has highlighted the aggravating role of exposure to NSAIDs on bacterial infections in adults, based on the usual septic severity Levy's score (SSS), and mortality, but it delays adequate antibiotics (Legras, Critical Care, 2009)
* Community-acquired bacterial infections in adults exposed to NSAIDs are serious by their spread (multiple locations), and suppurative character requiring frequent use of invasive procedures such as surgery or drainage. The SSS does not reflect the seriousness of these infections. They are frequently associated with use of ibuprofen (63.4%), and self-medication practices (65.5%).

The main hypothesis is that NSAIDs exposure is associated with a specific severity of community-acquired bacterial infection, marked by dissemination, suppurative complications or even invasive procedures requirement.

Our objectives are also to:

* Describe what NSAID use terms are associated to the risk of serious bacterial infections: molecule, dosage, duration of exposure, access (prescription or self-medication), associated drugs.
* To determine what type (s) (s) of bacterial infection is worsened by exposure to NSAIDs.
* To determine if other risk factors contribute to severity of bacterial community acquired infection
* To describe hospital costs associated to such severity of bacterial infection

ELIGIBILITY:
Inclusion Criteria:

* Patient : adult patient hospitalized in managed care organization (MCO) in one of the study centers for severe community bacterial infection, infected with more than one site, and / or abscess collection, and / or a per-cutaneous drainage of the infection, and / or septic surgery
* Control: Patient hospitalized in the same center (different service or not), during the week or months of the inclusion of cases for infection without abscess or invasive procedure, only one infected site

Exclusion Criteria:

* Hematologic or solid neoplasia undergoing chemotherapy, long-term corticosteroid, chronic exposure to NSAIDs, ongoing treatment with methotrexate or monoclonal antibody (anti-tumor necrosis factor (ant-TNF) particular), chronic buffy neutropenia, surgical site infections, catheter infections, disorders of consciousness or cognitive neuro-against-indicating the administration of the drug exposure questionnaire adults under guardianship, minor, no insurance disease, patients already included in a biomedical research with taking medication blind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arm type: patient Arm description: adult patient hospitalized in MCO in one of the study centers for severe community bacterial infection, infected with more than one site, and / or abscess collection, and / or a per-cutaneous drainage of the infection, and / or septic surgery.
  Arm type: control Arm description: Patient hospitalized in the same center (different service or not), during the week or months of the inclusion of cases for infection without abscess or invasive procedure, only one infected site Pairing criteria (case/control analysis): age/Charlson score/type of infection/centre
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
exposure to NSAIDs | From the inclusion (J0) to the the end of hospital stay, up to three months
  The risk studied is the exposure to NSAIDs, the overall medication history will be collected for cases and controls. The standard questionnaire to document medications history, including self-medication, was previously published (Asseray et al., 2013) The window of exposure to drugs is defined as 14 days before hospital admission. Drug exposure will be assessed at the time of inclusion.

SECONDARY OUTCOMES:
Name of NSAIDS | 36 months
  Describe what NSAIDs terms of use contribute to the risk of serious bacterial infections
type of bacterial infection at risk of worsening when exposed to NSAIDs | 36 months
  Describe what type of bacterial infection is at risk of worsening when exposed to NSAIDs.
other drugs exposure assessed by questionnaire | 36 months
Duration of NSAID exposure | 36 months
self-medication assessment | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Epaulard, PU-PH, Principal Investigator — University Hospital, Grenoble; Eric DENES, PH, Principal Investigator — University Hospital, Limoges; Thomas Guimard, PH, Principal Investigator — LA ROCHE SUR YON HOSPITAL; Louis BENARD, PU-PH, Principal Investigator — Tours University Hospital; Thierry MAY, PU-PH, Principal Investigator — Central Hospital, Nancy, France; Annie-Pierre JONVILLE-BERA, PH, Principal Investigator — Tours University Hospital

IPD SHARING:
Plan to Share IPD: No